CLINICAL TRIAL: NCT02432339
Title: Comparing the Effects of an Immunosuppressant (Mycophenolate Mofetil or MMF) on the Urinary Sodium Excretion Response to Mental Stress in a Crossover Design (MMF)
Brief Title: Effects of an Immunosuppressant Mycophenolate Mofetil or MMF on the Urinary Sodium Excretion Response to Mental Stress
Acronym: MMF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Gregory Harshfield, Director, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 611878
Record Dates: First submitted 2015-04-17; First posted 2015-05-04 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Psychological Stress; Hypertension, Renal
Keywords: immune system; RENIN-ANGIOTENSIN SYSTEM
MeSH Terms: conditions — Stress, Psychological; Hypertension, Renal | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mycophenolate mofetil (MMF) (Experimental): Mycophenolate Mofetil (MMF) 500 mg tablet twice a day for 7 1/2 days.
  Interventions: Drug: mycophenolate mofetil (MMF)
- Placebo (Placebo Comparator): Placebo (sugar pill) in the same size capsule that the MMF is used in - twice a day for 7 1/2 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mycophenolate mofetil (MMF) — an immunosuppressant - 500 mgs twice a day for 7 1/2 days - in capsule form
  Other Names: CellCept Chemical formula: C23H31NO7 Drugbank ID: DB00688
  Arms: mycophenolate mofetil (MMF)
Drug: Placebo — a sugar pill - 500 mgs twice a day for 7 1/2 days - in the same capsule form as the MMF
  Other Names: a sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if stopping the stress induced increase in inflammation will prevent sodium retention which in turn increases blood pressure. Each subject will test two separate times. One week, they will be taking a daily dose of mycophenolate mofetil (MMF), the other week they will be taking a placebo.

DETAILED DESCRIPTION:
This study will involve a screening visit and two testing weeks over an approximate 3 week period (this includes a one week "washout" period).

Each testing week will have a 3 day salt-controlled diet prior to testing and an approximate 3-hour testing period on Day 4. The 3-hour testing period will include 10 minutes of a baseline rest, 45 minutes of mild stress (competitive video game), and 45 minutes of a recovery rest. A total of 4 blood and 4 urine samples will be collected during the 3-hour period. Each blood draw will consist of about 7 teaspoons for a total of 28 teaspoons per testing week.

During the screening and testing, I will be asked to take the MoCA (the Montreal Cognitive Assessment) test in order to measure cognitive thinking after stress. It is a brief 30-question test which takes around 10 minutes to complete. It measures different types of cognitive abilities, including orientation (the approximate position of something/someone), short-term memory (remember information for a short period of time), executive function (planning and problem solving), language abilities (assign appropriate names to appropriate items), and visuospatial ability (determine distance from one object to another). Each question is awarded a particular number of points depending on the accuracy of the answers given. We will be looking to see if the total number of points earned changes in response before and after stress.

Screening Visit: I will come to the GPI or the CRU for a screening visit that will last about 90 minutes. The study will be described in detail and an informed consent will be obtained. Vital signs will be taken (blood pressure, height, weight and BMI - Body Mass Index. A health history and a limited physical exam will be conducted by Dr. White (or a physician delegate) to insure that it is safe for me to participate in the study. A blood sample will be obtained from me to make sure nothing is wrong with my kidneys or liver or have any other chronic illness. If all lab work returns with no abnormalities, then I will be cleared to participate in one of the crossover studies.

I will also select my food and drink items from a food menu for the 3-day diet prior to testing. The items I select will give me enough to eat and drink for the 3 days. All food and drink items will be packed in coolers that I will be responsible for picking up and dropping off daily. I am not to eat any food or drink item(s) other than those provided, except for water. To make sure that I am following the diet, I will be asked to return all of my food wrappers and drink containers to the GPI or CRU. I will also be asked to collect an overnight urine sample each night so that they can see how much salt I am taking in each day. My testing weeks will also be scheduled at this visit.

The last thing that I will be asked to do for the screening visit, is to take the MoCA test which will take approximately 10 minutes. Someone from the research team will instruct me as to what to do for each question and I will answer each one to the best of my ability.

Testing Week One: The week prior to my scheduled testing week, I will pick up my food coolers for the 3 day study diet along with my 7 ½ day prescription of either the MMF or the placebo. In addition, if I am female, I will have to give a urine sample so that a pregnancy test can be performed to make sure I am not pregnant before I start taking the medication. Should the pregnancy test show positive, I will not be allowed to continue participating in the study. I will take the study medication (either MMF or a placebo) 500 mgs twice a day for the 71/2 days as instructed, taking my last dose the morning of testing at GPI.

The coolers will contain the food and drink items that I selected previously at my screening visit. I will also receive the overnight urine collection bottles. During the diet phase of testing, I will collect a urine sample before I go to bed each night and record the time (write the time on the bottle). I will also collect a urine sample as soon as I wake up each morning and record the time. I will be returning the urine collection bottles and food coolers to GPI or CRU starting on the second day of the diet phase. This means that I will return my Monday cooler and urine collection bottle on Tuesday (Day 2). I will then return my Tuesday cooler and collection bottle on Wednesday (Day 3). On Thursday (testing day), I will bring back my Wednesday cooler and urine collection bottle. During the diet phase of the study, if I am female, a pregnancy test will be performed on each overnight urine sample to ensure that I am not pregnant.

On testing day, I will bring with me my Wednesday cooler and overnight urine sample and will be given breakfast before testing begins. Again, if I am female, a pregnancy test will be performed on my last (Wednesday) overnight urine sample to ensure I am not pregnant. I will be taken to a private room for testing and placed into a comfortable reclining chair. A nurse/phlebotomist will insert a small needle attached to a plastic tube called a catheter into a vein in my hand or arm. This procedure will allow the nurse/phlebotomist to collect the 4 blood samples over the 3-hour testing period. The needle stick may cause some temporary pain and may result in a black and blue mark. A device that automatically takes blood pressure will then be put on the opposite arm. I will also be given water in order to take my last dose of medication before testing begins and to sip on during the duration of testing. During the first 10 minute baseline rest period, I will relax in a reclining chair. I can listen to music, read a book or magazine or watch movies to pass the time. My blood pressure will be taken before and after this 10 minute rest period. Once the baseline rest period is over, a blood and urine sample will be collected.

During the stress period, I will play a video game against another subject for 45 minutes. My blood pressure will continue to be measured every 10 minutes. I will also continue to sip on water during this time. At the end of the game, another blood and urine sample will be collected. I will then be asked to complete the MoCA test a second time. It will be the same questions I was asked during the screening visit. A research team member will instruct me again as to how to answer each question and I will answer them to the best of my ability.

The last 45 minute recovery period of relaxation will be the same as the first (reading, listening to music or watching movies). My blood pressure will continue to be taken every 10 minutes. Once the 45 minutes has ended the last blood and urine sample will be collected and the testing day will then be completed.

Testing Week Two: The procedures for the Testing Week 2 are the same as Week 1. I will be on the controlled salt diet for 3-days, will take the study medication twice a day and will do the 3-hour testing on the 4th day. Like the first week, there will be 10 minute baseline rest period, 45 minutes stress period of the competitive video game and 45 minutes recovery rest period. Blood and urine samples will also be collected and I will be asked to take the MoCA test just like during Week 1 testing. Approximately 56 teaspoons of blood will be collected during the entire study. This blood will be used to examine how biochemical factors (stress hormones) relate to blood pressure and cardiovascular (heart) health. The DNA (genetic material) from the blood will be studied for genes relating to high blood pressure and other genes that may be related to the risk of cardiovascular disease. The blood, urine and DNA samples may be stored and used for other similar studies by Dr. Harshfield, Dr. Harris and Dr. Dong. The genetic results from these studies will not be told to myself and will not be given to any doctor or other individual.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Not pregnant or breastfeeding
* Does not have high blood pressure
* Currently not taking any medications that may effect blood pressure

Exclusion Criteria:

* Pregnant or breastfeeding
* Has High Blood pressure
* Taking medication that may effect blood pressure
* Failed Screening blood sample lab results - reviewed by study designated doctor

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04-22 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Urinary sodium excretion rate | 2 hours
  primary variable of interest is the difference in stress induced changes in sodium excretion between placebo and treatment conditions.

SECONDARY OUTCOMES:
Hemodynamics- change in systolic blood pressure compared to changes in sodium excretion | 2 hours
  measures of change in systolic blood pressure compared to changes in sodium excretion in treatment verses placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Harshfield, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The following avenues of dissemination will be used to share the research results:
  Publications: Study results that are published will be made available in PubMed-cited journals and submitted to PubMed Central in a timely fashion. All data that involves human subjects will be de-identified and presented in a format that protects the identity and privacy of study participants. Publication of results in professional peer reviewed journals will be a priority. All publications will acknowledge the support of the NIH/NHLBI per notice of award guidelines. Every effort will be made to publish scientific results from this project in a timely manner.
  Presentation at Scientific meetings: Abstracts will be submitted to the local, regional, and national association meetings such as annual meetings of the American Heart Association Council for High Blood Pressure Research, American Society of Hypertension, and American Society of Nephrology as well as Experimental Biology.
Supporting Information: Study Protocol